CLINICAL TRIAL: NCT01480323
Title: A Phase II Study to Evaluate Safety and Efficacy of Combined Treatment With Ipilimumab and Intratumoral Interleukin-2 in Pretreated Patients With Stage IV Melanoma
Brief Title: A Phase II Study to Evaluate Safety and Efficacy of Combined Treatment With Ipilimumab and Intratumoral Interleukin-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Benjamin Weide, M.D., Dr. Benjamin Weide, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5027000
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Malignant Melanoma
Keywords: Malignant melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; aldesleukin; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab (Experimental): Ipilimumab i.v. + Interleukin-2 intratumoral
  Interventions: Drug: Interleukin-2; Drug: Ipilimumab

INTERVENTIONS:
Drug: Interleukin-2 — intratumoral injections of 9 MIU/day on days 1, 4, 8, 11, 15, 18, 22 and 25. The administered dose will be distributed between all injectable soft-tissue metastases
  Other Names: Proleukin®
Drug: Ipilimumab — IV infusion, 3 mg/kg, day 2, 23, 44, 65
  Other Names: Proleukin

SUMMARY:
The current clinical trial shall clarify a synergistic effect with regards to efficiency by the combination of intratumoral injection of interleukin-2 (IL-2) and the intra-venous application of ipilimumab.

DETAILED DESCRIPTION:
Intratumoral injection of interleukin-2 (IL-2) into melanoma metastases is a highly efficient local treatment. Furthermore, a systemic effect is assumed based on the observation of a favorable long term outcome. However, objective responses in untreated lesions have not been observed yet. Ipilimumab seems to be efficient in a subset of treated patients by inhibition of down-regulation of tumor-specific cellular immune-responses. In the context of the proposed trial, we assume (i) that ipilimumab could potentiate systemic melanoma-specific immune responses, which are primarily induced by intratumoral IL-2 and (ii) that these immune responses become more effective with regards to not IL-2 injected distant lesions. Therefore we assume a synergistic effect with regards to efficiency by the combination.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent;
* Histological diagnosis of malignant melanoma;
* Stage IV melanoma;
* At least one injectable lesions > 5 mm (longest diameter) or at least 5 injectable lesions < 5 mm.
* Measurable disease. Note: lesions, which are designated for direct IL -2 injections, must not be considered in the evaluation of measurability;
* Men and women, at least 18 years of age;
* Patient must have demonstrated 1 of the following in response to at least 1 cycle of 1 or more systemic regimens:

  1. relapse following an objective response (PR/CR);
  2. failed to demonstrate an objective response (PR/CR); or
  3. inability to tolerate treatment due to unacceptable toxicity
* At least 4 weeks since treatment (chemotherapy, biochemotherapy, surgery, radiation, immunotherapy, etc.) for melanoma and recovered from any clinically significant toxicity experienced during treatment;
* Life expectancy ≥3 months;
* ECOG performance status of 0 or 1;
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab;
* No known active or chronic infection with HIV, Hepatitis B, or Hepatitis C
* Required values for initial laboratory tests:
* Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study and for up to 26 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized

Exclusion Criteria:

* Any other prior malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix;
* Ocular melanoma; mucosal melanoma
* Either untreated or symptomatic central nervous system (CNS) metastases (patients with brain metastases who are identified at screening may be rescreened after the lesion(s) have been appropriately treated);
* Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome). Patients with vitiligo may be included.
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* A history of prior systemic treatment with ipilimumab, CD137 agonist, CTLA 4 inhibitor, CTLA-4 agonist or IL-2 in stage IV melanoma.
* Concomitant or less than 4 weeks off therapy with any of the following: interferon; other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; chronic use of systemic corticosteroids.
* Women of childbearing potential (WOCBP), defined in Section 5.3, who:

  1. are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 26 weeks after cessation of study drug, or
  2. have a positive pregnancy test at baseline, or
  3. are pregnant or breastfeeding.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Control rate | at week 12
  To determine efficacy of the combined treatment with ipilimumab and intratumoral IL-2 by assessment of Disease control rate according to immune-related response criteria (irDCR) at week 12

SECONDARY OUTCOMES:
Tolerability | within 12 months after start of treatment
  Tolerability according to NCI-CTCAE-Criteria (version 4)
Overall survival | within 12 months after start of treatment
  Overall survival
Best Overall Response Rate | within 12 months after start of treatment
  Best Overall Response Rate (irBORR) according to irRC
Overall response rate | at week 12
  Overall response rate (sum of irPR and irCR) according to irRC
Overall Response Rate | at week 12
  Overall Response Rate according to modified mWHO criteria
Best Overall Response Rate | within 12 months after start of treatment
  Best Overall Response Rate according to modified mWHO criteria
Response rate of injected metastases only | at week 12
  Response rate of injected metastases only
Rate of patients with substantial increase of anti-melanoma T-cells in peripheral blood during treatment | within 22 weeks after start of treatment
  Rate of patients with substantial increase of anti-melanoma T-cells in peripheral blood during treatment
Changes in T-cell subsets during treatment | within 22 weeks after start of treatment
  Changes in T-cell subsets during treatment
Changes in subsets of tumor-infiltrating lymphocytes during treatment | within 22 weeks after start of treatment
  Changes in subsets of tumor-infiltrating lymphocytes during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Weide, Dr. med., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany